CLINICAL TRIAL: NCT00597363
Title: Neptune Pad ® Compared to Conventional Manual Compression for Access Site Management After Peripheral Percutaneous Transluminal Procedures
Brief Title: Neptune Pad ® Compared to Conventional Manual Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna General Hospital (Other)
Responsible Party: Prof.Dr. Wolfgang Mlekusch, Department of Internal Medicine, Division of clinical Angiology, MUW Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EK 433/2004
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Postoperative Hemorrhage
Keywords: vascular access site; arterial puncture; femoral pseudoaneurysm
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Neptune PAD utilization to accelerate closure of the vascular access site
  Interventions: Device: Neptune P.A.D. (R)
- 2 (Active Comparator): manual compression for closure of the vascular access site
  Interventions: Other: conventional manual compression

INTERVENTIONS:
Device: Neptune P.A.D. (R) — The Neptune Pad ® (Biotronik GmbH & Co. KG, Berlin, Germany) is a soft and hydrophilic wound dressing, which has been developed to accelerate local hemostasis, reduce compression times, enable early ambulation and minimize the risk for bleeding complications. Neptune Pad ® consists of calcium alginate, which is cationically charged and exerts potent procoagulant properties.
  Arms: 1
Other: conventional manual compression — The most common technique for puncture site management is manual compression. This technique requires an extended pressure on the puncture site, and after achievement of hemostasis a pressure bandage is applied for several hours at bed rest.
  Arms: 2

SUMMARY:
BACKGROUND. Arterial access site complications remain the most frequent adverse events after percutaneous transluminal procedures. We investigated the safety and efficacy of the pro-coagulant wound dressing Neptune Pad ® compared to conventional manual compression for access site management after peripheral percutaneous interventions.

METHODS. We enrolled 201 consecutive patients and randomly assigned patients for Neptune Pad ® (n=100) vs. conventional manual compression (n=101). Patients were followed clinically until hospital discharge and by duplex ultrasound at 24 hours postprocedure for occurrence of access site complications. Time-to-hemostasis and time-to-ambulation were recorded, patients´ and physicians´ discomfort were measured using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* All inguinal punctures (common femoral, superficial femoral and deep femoral artery, antegrade and retrograde access) were included.
* No specific limitations of anti-platelet or anti-coagulant medication were specified.

Exclusion Criteria:

* Patients with extreme obesity (BMI above 35 kg/m2) were not included according to the manufactures' recommendations.
* Furthermore, patients with known hypersensitivity to components of the device were not eligible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schillinger, MD, Principal Investigator — Professor
Locations (1):
- General Hospital Vienna, Vienna, Austria

REFERENCES:
- [Background] Mlekusch W, Dick P, Haumer M, Sabeti S, Minar E, Schillinger M. Arterial puncture site management after percutaneous transluminal procedures using a hemostatic wound dressing (Clo-Sur P.A.D.) versus conventional manual compression: a randomized controlled trial. J Endovasc Ther. 2006 Feb;13(1):23-31. doi: 10.1583/05-1679.1. PMID 16445320